CLINICAL TRIAL: NCT01577862
Title: Randomised, Open-Label Clinical Trial on The Efficacy of Colistin Plus Rifampicin Treatment Versus Colistin Alone for Severe Infections Due to Multidrug-Resistant Acinetobacter Baumannii
Brief Title: Colistin and Rifampicin for MDR-Acinetobacter
Acronym: CoRAb
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Federico II University (Other)
Responsible Party: Principal Investigator, Riccardo Utili, Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM7X9F8K
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Infection Due to Resistant Bacteria; Pneumonia, Ventilator-Associated; Hospital Acquired Pneumonia; Infection of Bloodstream; Infectious Disease of Abdomen
Keywords: ACINETOBACTER BAUMANNII; COLISTIN; RIFAMPICIN; THERAPY; RESISTANCE
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Sepsis; Intraabdominal Infections | interventions — Colistin; colistinmethanesulfonic acid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colistin (Active Comparator): Colistin alone, 2 million units every 8 hours intravenously or according to renal function
  Interventions: Drug: Colistin
- Colistin plus Rifampicin (Experimental): Colistin, 2 million units every 8 hours intravenously or according to renal function, plus Rifampicin, 600 mg every 12 hours intravenously
  Interventions: Drug: Colistin; Drug: Rifampicin

INTERVENTIONS:
Drug: Colistin — 2 million units every 8 hours intravenously for at least 10 and up to a maximum of 21 days
  Other Names: Sodium colistimethate
Drug: Rifampicin — 600 mg every 12 hours intravenously
  Other Names: Rifampin
  Arms: Colistin plus Rifampicin

SUMMARY:
Acinetobacter baumannii causes severe infections (pneumonia, bacteremia, organ space) with high lethality in hospitalised critically ill patients. It can acquire resistance to all classes of antibiotics (multidrug resistance, MDR) except an 'old' drug, colistin, which may be the only therapeutic option. However, colistin is not registered for this indication. The addition of rifampicin to colistin has been shown to be synergistic in vitro, and may be promising in vivo, but this combination has not been studied in comparison with colistin alone.

The purpose of this randomised, open-label, multicentre clinical trial is to assess whether the association of colistin and rifampicin reduces significantly the mortality of patients with severe MDR A. baumannii infections compared with colistin alone.

The trial will enroll 210 patients from intensive care units (ICU) of five tertiary care hospitals where MDR A. baumannii infection is endemic with epidemic phases. Patients will be randomly allocated to either colistin alone (control arm) or colistin plus rifampicin (experimental arm).

Primary end point is overall mortality, defined as death occurring within 30 days from randomisation.

Secondary end points will be disease-specific death, microbiological eradication, hospitalization length, emergence of resistance to colistin during treatment.

DETAILED DESCRIPTION:
This study is designed as a multicentre open-label, parallel randomised, controlled trial. Patients will be randomly allocated to two treatment arms: 1) colistin alone (control arm); 2) colistin, plus rifampicin (experimental arm). The study will be carried out over 2 years according to the principles of good clinical practice.

The study population is represented by adult hospitalised patients with severe nosocomial infections due to multi-drug resistant A. baumannii, susceptible to colistin. It will be performed in intensive or sub-intensive care units of 5 Italian clinical centres where MDR A. baumannii infection is endemic with epidemic phases. All adult subjects, irrespective of age, will be included in the study, thus also elderly subjects will be eligible. Large eligibility criteria are warranted by the pragmatic approach of the study, the severe prognosis of these patients and the lack of effective alternative treatments.

Enrollment procedure: At the time of A. baumannii isolation, inclusion and exclusion criteria will be checked by the pertinent centre.

Once obtained the informed consent, subjects will be randomized to treatment. No patient may be enrolled in a centre before the formal approval of the Ethics Committee of that Institution.

Accrual time: according to the sample size estimate (see below) and based on the current incidence of MDR A. baumannii severe infections of 12-14 cases per month in the five participating centres, the accrual time will last approximately 18 months to achieve the planned sample size.

Severe infections include hospital acquired pneumonia (HAP), ventilator associated pneumonia (VAP), bloodstream infection, intra-abdominal infection or other organ-space infections.

Multi-drug resistant A. baumannii is defined as clinical isolates resistant to carbapenems and to all other antimicrobial drug classes, except colistin, irrespective of rifampicin activity.

Severity of illness is assessed by the SAPS II score. This will be considered low or high according to a SAPS II score below/equal to or higher than 40, respectively.

Patients will be randomly allocated into two treatment arms: 1) colistin alone, 2 million units every 8 hours intravenously or according to renal function (control arm); 2) colistin, 2 million units every 8 hours intravenously or according to renal function, plus rifampicin, 600 mg every 12 hours intravenously (experimental arm).

Treatment will be administered for at least 10 days and up to a maximum of 21 days. Duration of treatment will be established by the physician in charge. The end of treatment (EoT) evaluation will be performed the day of treatment discontinuation. The end of study (EoS) (follow-up) evaluation will be performed 30 days after randomization.

Treatment will be discontinued in the following instances: clinical cure with or without microbiological eradication; occurrence of significant renal or liver toxicity; patient death. Throughout the study, patients will receive routine intensive care support by the physician in charge according to standard diagnostic and therapeutic guidelines.

Clinical cure is defined by disappearance of symptoms and signs of infection, irrespective of A. baumannii eradication at the site of infection. Therapeutic failure is defined as worsening or no improvement of clinical conditions on therapy with persistently positive A. baumannii cultures.

Renal and liver function will be monitored by daily measurements of creatinine, aminotransferase and direct bilirubin serum levels.

Drug dosages will be adjusted according to renal and liver function. Renal toxicity is defined as decrease of creatinine clearance below 50 ml/min or >50% reduction in the creatinine clearance relative to the baseline. Hepatic toxicity is defined as increase of direct bilirubin above 3 mg/dl.

Surveillance cultures from the original source of isolation (blood, bronchial aspirate, urines or drainage fluids) will be obtained on admission and repeated weekly, or whenever clinically needed, during and after treatment to monitor persistence versus eradication of A. baumannii at the infected site. In vitro activity of colistin and rifampicin will be checked against all A. baumannii repeat isolates to detect development of resistance. Identification and antibiotic susceptibility of A. baumannii isolates will be performed at each centre using an automated system. Species identification will be confirmed by molecular biology.

ELIGIBILITY:
Inclusion Criteria:

* clinical and microbiological evidence of a severe infection due to multi-drug resistant A. baumannii during hospitalization
* susceptibility of the A. baumannii isolate to colistin (MIC < or =2 mg/l).

Exclusion Criteria:

* age below 18 years
* treatment with one of the study drugs prior to the diagnosis of A. baumannii infection
* severe liver dysfunction
* history of prior hypersensitivity to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 day
  The study primary outcome is patient overall mortality, defined as death occurring during hospitalisation or within 30 days from randomization.

SECONDARY OUTCOMES:
Disease-specific death | 30 days after randomization
  Disease-specific death or A. baumannii infection-related death is defined as death occurring in the presence of persistent signs and symptoms of A. baumannii infection (persistent pneumonia, septic shock) and/or when it occurs within the first week of antibiotic treatment without any other clear explanation.
Microbiological eradication | 30 day
  Microbiological eradication is defined as the disappearance of A. baumannii in cultures from blood, bronchial aspirate, urines and drainage fluids.
Hospitalization length | From admission to hospital discharge, an average of 30 days
  Hospitalization length is calculated as days in the hospital as well as days in the intensive care unit since diagnosis of A. baumannii infection.
Emergence of resistance to colistin | From day 1 to the end of study evaluation, 30 days after randomization
  Emergence of resistance is defined as the detection during treatment of an A. baumannii isolate showing resistance to colistin (MIC >2 mg/l).
Toxicity | From day 1 to the end of treatment evaluation, performed between day 10 and day 21
  Renal toxicity is defined as decrease of creatinine clearance below 50 ml/min or >50% reduction in the creatinine clearance relative to the baseline. Hepatic toxicity is defined as increase of direct bilirubin above 3 mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Utili, MD, Principal Investigator — University of Campania Luigi Vanvitelli

REFERENCES:
- [Derived] Durante-Mangoni E, Signoriello G, Andini R, Mattei A, De Cristoforo M, Murino P, Bassetti M, Malacarne P, Petrosillo N, Galdieri N, Mocavero P, Corcione A, Viscoli C, Zarrilli R, Gallo C, Utili R. Colistin and rifampicin compared with colistin alone for the treatment of serious infections due to extensively drug-resistant Acinetobacter baumannii: a multicenter, randomized clinical trial. Clin Infect Dis. 2013 Aug;57(3):349-58. doi: 10.1093/cid/cit253. Epub 2013 Apr 24. PMID 23616495